CLINICAL TRIAL: NCT02164864
Title: A Prospective Randomised, Open Label, Blinded Endpoint (PROBE) Study to Evaluate DUAL Antithrombotic Therapy With Dabigatran Etexilate (110mg and 150mg b.i.d.) Plus Clopidogrel or Ticagrelor vs. Triple Therapy Strategy With Warfarin (INR 2.0 - 3.0) Plus Clopidogrel or Ticagrelor and Aspirin in Patients With Non Valvular Atrial Fibrillation (NVAF) That Have Undergone a Percutaneous Coronary Intervention (PCI) With Stenting
Brief Title: Evaluation of Dual Therapy With Dabigatran vs. Triple Therapy With Warfarin in Patients With AF That Undergo a PCI With Stenting (REDUAL-PCI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1160.186; 2013-003201-26 (EudraCT Number)
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Percutaneous Coronary Intervention
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran; Warfarin; Aspirin; Clopidogrel; Ticagrelor

ARMS (3):
- Dabigatran Etexilate 110mg (Experimental): Patient to receive Dabigatran Etexilate 110mg twice a day (BID)
  Interventions: Drug: Dabigatran Etexilate 110mg; Drug: Clopidogrel or Ticagrelor
- Dabigatran Etexilate 150mg (Experimental): Patient to receive Dabigatran Etexilate 150mg twice a day (BID)
  Interventions: Drug: Dabigatran Etexilate 150mg; Drug: Clopidogrel or Ticagrelor
- Warfarin (Active Comparator): Warfarin doses to maintain INR
  Interventions: Drug: Warfarin 3mg; Drug: Aspirin; Drug: Clopidogrel or Ticagrelor; Drug: Warfarin 5mg; Drug: Warfarin 1mg

INTERVENTIONS:
Drug: Dabigatran Etexilate 110mg — Active treatment
  Arms: Dabigatran Etexilate 110mg
Drug: Warfarin 3mg — Active comparator
  Arms: Warfarin
Drug: Aspirin — Active comparator
  Arms: Warfarin
Drug: Dabigatran Etexilate 150mg — Active treatment
  Arms: Dabigatran Etexilate 150mg
Drug: Clopidogrel or Ticagrelor — Active comparator
  Arms: Warfarin
Drug: Clopidogrel or Ticagrelor — Active comparator
  Arms: Dabigatran Etexilate 110mg
Drug: Warfarin 5mg — Active comparator
  Arms: Warfarin
Drug: Clopidogrel or Ticagrelor — Active comparator
  Arms: Dabigatran Etexilate 150mg
Drug: Warfarin 1mg — Active comparator
  Arms: Warfarin

SUMMARY:
The main objective of this study is to compare a Dual Antithrombotic Therapy (DAT) regimen of 110mg dabigatran etexilate b.i.d. plus clopidogrel or ticagrelor (110mg dabigatran etexilate (DE) DAT) and 150mg dabigatran etexilate b.i.d. plus clopidogrel or ticagrelor (150mg DE-DAT) with a Triple Antithrombotic Therapy (TAT) combination of warfarin plus clopidogrel or ticagrelor plus Aspirin (ASA) <= 100mg once daily (warfarin-TAT) in patients with Atrial Fibrillation that undergo a PCI with stenting (elective or due to an Acute Coronary Syndrome).

The study aims to show non-inferiority of each dose of DE-DAT when compared to Warfarin-TAT in terms of safety. Safety will be determined by comparing the rates of bleeding events, assessed using the modified International Society of Thrombosis and Haemostasis classification of Major Bleeding and Clinically Relevant Non Major Bleeding Events.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients aged >=18 years
* Patients with Non Valvular Atrial Fibrillation
* Patient presenting with:

An Acute Coronary Syndrome (ACS) (ST elevation myocardial infarction (STEMI), NonSTEMI [NSTEMI] or unstable angina [UA]) that was successfully treated by PCI and stenting (either Bare Metal Stent (BMS) or Drug Eluting Stent) Or Stable Coronary Artery Disease with at least one lesion eligible for PCI that was successfully treated by elective PCI and stenting (either BMS or DES)

* The patient must be able to give informed consent in accordance with International Conference on Harmonisation Good Clinical Practice guidelines and local legislation and/or regulations.

Exclusion criteria:

* Patients with a mechanical or biological heart valve prosthesis
* Cardiogenic shock during current hospitalisation
* Stroke within 1 month prior to screening visit
* Patients who have had major surgery within the month prior to screening
* Gastrointestinal haemorrhage within one month prior to screening, unless, in the opinion of the Investigator, the cause has been permanently eliminated
* Major bleeding episode including life-threatening bleeding episode in one month prior to screening visit
* Anaemia (haemoglobin <10g/dL) or thrombocytopenia including heparin-induced thrombocytopenia (platelet count <100 x 109/L) at screening
* Severe renal impairment (estimated Creatinine Clearance (CrCl) calculated by Cockcroft-Gault equation) <30mL/min at screening
* Active liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2725 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (418):
- United States (45):
  - Cardiology P.C., Birmingham, Alabama
  - Verde Valley Medical Center, Cottonwood, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Arkansas Cardiology, PA, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - Aurora Denver Cardiology Associates, PC, Aurora, Colorado
  - University of Florida College of Medicine, Jacksonville, Florida
  - Watson Clinic, LLP, Lakeland, Florida
  - Community Clinical Research Center, Anderson, Indiana
  - Midwest Cardiovascular Research and Education Foundation, Elkhart, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - Richmond Cardiology Associates Research, LLC, Richmond, Indiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Maine Medical Center, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Cape Cod Research Institute, Hyannis, Massachusetts
  - Mid Michigan Medical Center, Midland, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Saint Mary's Medical Center dba Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - Kansas City Veterans Administration Medical Center, Kansas City, Missouri
  - Saint Anthony's Medical Center, St Louis, Missouri
  - St. Michaels Medical Center, Newark, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - VA Western New York Healthcare System, Buffalo, New York
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Altru Health System, Grand Forks, North Dakota
  - Cardiovascular Research Center, Toledo, Ohio
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Pinnacle Health Harrisburg Hospital, Harrisburg, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Chattanooga Heart Institute, Chattanooga, Tennessee
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Scott and White Healthcare, Round Rock, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Wichita Falls Heart Clinic, Wichita Falls, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bayview Physicians Services PC dba Cardiovascular Associates, Virginia Beach, Virginia
  - Holy Family Memorial, Inc, Manitowoc, Wisconsin
- Argentina (9):
  - Fundación Favaloro, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Instituto Cardiovascular de Buenos Aires, CABA
  - Consultorios Asociados de Endocrinología e Invest Clínica, Capital Federal
  - Instituto de Cardiología de Corrientes, Corrientes
  - Sanatorio Allende, Córdoba
  - Instituto CER, Quilmes
  - Inst.Cardiovascular San Luis, San Luis
  - Investigaciones Clinicas Tucumán, San Miguel de Tucumán
- Australia (8):
  - Pendlebury Research, Adamstown, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Heartcare Victoria, Bundoora, Victoria
  - The Geelong Hospital, Geelong, Victoria
- Austria (3):
  - Order Hospital Elisabethinen Linz, Linz
  - LKH Salzburg, Univ. Clinic, Salzburg
  - Wilhelminenspital, Vienna
- Belgium (10):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - Bonheiden - HOSP Imelda, Bonheiden
  - Brussels-UNIV Brugmann -Horta, Brussels
  - Brussels - UNIV UZ Brussel, Brussels
  - AZ Sint-Lucas - Campus Sint Lucas, Ghent
  - Charleroi - HOSP St-Joseph, Gilly
  - Ziekenhuis Netwerk Antwerpen (ZNA) - Campus Middelheim, Middelheim
  - Sint-Niklaas - HOSP AZ Nikolaas (Campus St-Niklaas), Sint-Niklaas
  - Tienen - PRAC De Wolf, Axel, Tienen
  - Brussels - HOSP Europe (Ste-Elisabeth), Uccle
- Brazil (8):
  - Hospital Santa Isabel, Blumenau
  - Irmandade da Santa Casa de Misericordia de Curitiba, Campina Grande do Sul
  - Instituto de Cardiologia Rio Grande do Sul, Porto Alegre
  - Hospital de Base - Fac Med de Sao Jose do Rio Preto, São José do Rio Preto
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital Sao Paulo - UNIFESP, São Paulo
  - INCOR e Hospital das Clínicas da Universidade de São Paulo, São Paulo
  - Eurolatino pesquisas Médicas Ltda, Uberlândia
- Bulgaria (6):
  - MHAT "Deva Maria", Dept. of Cardiology, Burgas, Burgas
  - SHAT in Cardiology EAD, Pleven, Pleven
  - MHAT"Sv.Georgi",Cardi.Clin., Plovdiv
  - MHAT "Sv. Vrach" EOOD, Cardiology Dept., Sandanski, Sandanski
  - City Clin.Univ.MPHAT EOOD,Clin.of Cardiology, Sofia, Sofia
  - Specialized Hosp.f.Active Treatment, Cardiology Dept, Yambol, Yambol
- Canada (11):
  - Calgary Heart Centre, Calgary, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Dr. R. Labonte Prof. Med. Corp, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - CHUS Fleurimont, Sherbrooke, Quebec
  - IUCPQ (Laval University), Ste-Foy, Quebec
- Chile (4):
  - Hospital San Juan de Dios, Santiago
  - Centro de Estudios Clinicos Barros Luco, Santiago
  - Hospital Las Higueras, Talcahuano
  - CECMI Ltda, Temuco
- Colombia (6):
  - Fundación Clínica Abood Shaio, Bogotá
  - Fundación Santa Fe de Bogotá, Bogotá
  - Centro Médico Imbanaco de Cali S.A., Cali
  - Fundación Valle de Lili, Cali
  - Fundación Cardiovascular de Colombia, Floridablanca
  - Hospital Pablo Tobón Uribe, Medellín
- Croatia (5):
  - Clincal Hospital Centre Rijeka, Rijeka
  - Clinical Hosp.Merkur,Clin.Internal Med,Cardiology Dep,Zagreb, Zagreb
  - Clinical Hospital Sstre Milosrdnice, Cardiology Dept, Zagreb, Zagreb
  - University hospital center Zagreb, Zagreb
  - University Hospital Dubrava, Zagreb
- Czechia (12):
  - Amkardia, s.r.o. Brno, Brno
  - Hospital Jihlava, Jihlava
  - Karlovarska Reg.Hosp, Cardiology Dept, Karlovy Vary, Karlovy Vary
  - University Hospital Olomouc, Olomouc
  - Municipal Hospital Ostrava, Ostrava
  - General Faculty Hospital, Prague, Prague
  - Institute for Clinical and Experimental Medicine, Prague
  - University Hospital Motol, Prague
  - Hospital Slany, Internal Department, Slaný
  - Hospitals of Pardubice Region, Internal Department, Svitavy, Svitavy
  - Masaryk Hospital, Usti nad Labem, Ústí nad Labem
  - Hosp.of Pardubice Reg,Orlickoustecka,Internal Dept, Ustinad, Ústí nad Orlicí
- Aarhus Universitetshospital, Århus N, Denmark
- Finland (4):
  - HYKS, Kardiologian klinikka, Sydän- ja keuhkokeskus, Helsinki
  - StudyCor Oy, Jyväskylä
  - Keski-Pohjanmaan keskussairaala, Kardiologian pkl, Kokkola, Kokkola
  - TYKS, Turku
- France (12):
  - HOP Ambroise Paré, Boulogne-Billancourt
  - HOP de la Cavale Blanche, Brest
  - HOP Gabriel-Montpied, Clermont-Ferrand
  - HOP CHU de Grenoble, Grenoble
  - HOP St Joseph, Marseille
  - CLI du Pont de Chaume, Montauban
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Pasteur, Nice
  - HOP Lariboisière, Paris
  - HOP Salpêtrière, Cardio, Paris, Paris
  - CLI Saint-Hilaire, Rouen
  - HOP Rangueil, Toulouse
- Germany (47):
  - SLK-Kliniken Heilbronn GmbH, Bad Friedrichshall
  - Kerckhoff-Klinik, Bad Nauheim, Bad Nauheim
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen, Bad Oeynhausen
  - CIMS Studienzentrum Bamberg GmbH, Bamberg
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Charité - Universitätsmedizin Berlin, Berlin
  - Klinikum Bielefeld gGmbH, Bielefeld
  - St. Josef- und St. Elisabeth-Hospital gGmbH, Bochum
  - Universitätsklinikum Bonn AöR, Bonn
  - Allgemeines Krankenhaus, Celle, Celle
  - Klinikum Coburg gGmbH, Coburg
  - Helios Amper-Klinikum Dachau, Dachau
  - St. Johannes Hospital Dortmund, Dortmund
  - Städtisches Klinikum Dresden, Dresden
  - Praxisklinik Herz und Gefäße, Dresden
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Universitätsklinikum Frankfurt, Frankfurt
  - Städtisches Klinikum, Fulda, Fulda
  - Herz- und Gefäßzentrum (HGZ-Göttingen) am Krankenhaus Neu Bethlehem, Göttingen
  - Universitätsmedizin Göttingen, Georg-August-Universität, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Cardiologicum Hamburg, Hamburg
  - Westküstenkliniken Brunsbüttel und Heide gGmbH, Heide
  - HPK-Heidelberger Praxisklinik, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Asklepios Klinik Langen-Seligenstadt GmbH, Langen
  - Herzzentrum Leipzig GmbH, Leipzig
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Märkische Gesundheitsholding GmbH & Co. KG, Klinikum Lüdenscheid, Lüdenscheid
  - Universitätsklinikum Magdeburg AöR, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Carl-von-Basedow Klinikum Saalekreis gGmgH, Merseburg
  - Klinikum der Universität München - Campus Großhadern, München
  - Städtisches Klinikum München GmbH, München
  - Universitätsklinikum Münster, Münster
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Sana-Klinikum Remscheid GmbH, Remscheid
  - Universitätsmedizin Rostock, Rostock
  - Robert-Bosch-Krankenhaus GmbH, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Marien-Hospital-Wesel gGmbH, Wesel
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Greece (10):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Hippokration Hospital, Univ Clinic of Cardiology, Athens
  - General Hospital of Athens "Alexandra", Athens
  - General Hospital of Athens Konstantopoulio-Agia Olga, Athens
  - General Hospital of Attica "Sismanoglio - Amalia Fleming", Athens
  - General Hospital of Chios, Department of Cardiology, Chios
  - University General Hospital of Heraklion, Heraklion, Crete
  - Univ. Gen. Hosp. of Ioannina, Ioannina
  - University Hospital of Patras, Pátrai
  - University Hospital of Thessaloniki AHEPA, Thessaloniki
- Hong Kong (4):
  - Prince of Wales Hosp, Dept of Med & Therapeutics, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (7):
  - Gottsegen Gyorgy Hungarian Instit.of Cardiology,Budapest, Budapest
  - Semmelweis University, Budapest
  - Milit.Hosp.-State Health Cent., Budapest
  - University Debrecen Hospital, Debrecen
  - Bacs-Kiskun Megyei Onkormanyzat Hospital, Kecskemét
  - University of Pecs, Invasive Cardiology, Pécs
  - Univ. of Szeged, 2nd Dept. of Internal Med., Haematology, Szeged
- India (9):
  - Care Institute Of Medical Sciences, Ahmedabad
  - Medanta- The Medicity, Gūrgaon
  - Nizam's Institute of Medical Sciences, Hyderabad
  - B and M Patel Cardiac Centre, Shree Krishna Hospital,, Karamsad
  - Shri Krishna Hrudayalaya and Critical Care, Nagpur
  - Vijan Cardiac and Critical Care Centre, Nashik
  - Fortis Escorts Heart Institute, New Delhi
  - Byramjee Jeejeebhoy Medical College, Pune
  - King George's Hospital,, Seemandhra
- Ireland (4):
  - Mater Misericordiae University Hospital, Dublin
  - St James's Hospital, Dublin
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Hillel Yaffe Medical Center, Hadera, Hadera
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem 91031, Jerusalem
  - West.Galilee Med.Cent.Naharia, Nahariya
  - Rabin Medical Center Beilinson, Petah Tikva
- Italy (15):
  - Ospedale San Donato di Arezzo, Arezzo
  - ASST Papa Giovanni XXIII - A.O. Papa Giovanni XXIII, Bergamo
  - Fond. Poliambulanza Istituto, Brescia
  - A.O.U. Policlinico Vittorio Emanuele, Catania
  - Osp. Clin. SS. Anunziata, Chieti
  - Ospedale "Fabrizio Spaziani", Frosinone
  - Ospedale della Misericordia, Grosseto
  - Azienda Ospedaliera Vito Fazzi, Lecce
  - Osp. Pediatrico Aprano Pasquinucci, Massa
  - Ospedale Cardarelli, Napoli
  - Pol. Universitario Tor Vergata, Roma
  - Policlinico Gemelli, Roma
  - Presidio Ospedaliero di Saronno, Saronno (VA)
  - Ospedale Bolognini, Seriate
  - Ospedale Molinette, AO Città della Salute e della, Torino
- Japan (38):
  - Japanese Red Cross Nagoya Daini Hospital, Aichi, Nagoya
  - Hirosaki University Hospital, Aomori, Hirosaki
  - Chiba University Hospital, Chiba, Chiba
  - Kokura Memorial Hospital, Fukuoka, Kitakyushu
  - Fukuoka-Higashi Med. Ctr. Fukuoka, CV, Fukuoka, Koga
  - Shin Koga Hospital, Fukuoka, Kurume
  - Gumma Prefectural Cardiovascular Center, Gunma, Maebashi
  - National Hospital Organization Takasaki General Medical Center, Gunma, Takasaki
  - Fukuyama Cardiovascular Hospital, Hiroshima, Fukuyama
  - Tokeidai Memorial Hospital, Hokkaido, Sapporo
  - National Hospital Organization Hokkaido Medical Center, Hokkaido, Sapporo
  - Hyogo Brain and Heart Center, Hyogo, Himeji
  - The Veritas Hospital, Hyogo, Kawanishi
  - Kobe University Hospital, Hyogo, Kobe
  - Takahashi Hospital, Hyogo, Kobe
  - National Hospital Organization Kanazawa Medical Center, Ishikawa, Kanazawa
  - Iwate Medical University Hospital, Iwate, Morioka
  - Kagawa Prefectural Central Hospital, Kagawa, Takamatsu
  - Shonan Fujisawa Tokushukai Hospital, Kanagawa, Fujisawa
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Yokohama City Minato Red Cross Hospital, Kanagawa, Yokohama
  - Kyoto University Hospital, Kyoto, Kyoto
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Sakurabashi Watanabe Hospital, Osaka, Osaka
  - Osaka City Hospital Organization Osaka City General Hospital, Osaka, Osaka
  - Sayama General Clinic, Saitama, Sayama
  - National Hospital Organization Saitama National Hospital, Saitama, Wako
  - Kusatsu General Hospital, Shiga, Kusatsu
  - Omihachiman Community Medical Center, Shiga, Omihachiman
  - Tokushima Red Cross Hospital, Tokushima, Komatsushima
  - Nishiarai Heart Center Hospital, Tokyo, Adachi-ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-ku
  - Minamino Heart Clinic, Tokyo, Hachioji
  - Teikyo University Hospital, Tokyo, Itabashi-Ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-Ku
  - Itabashi Chuo Medical Center, Tokyo, Itabashi-Ku
  - Global Health and Medicine Ctr, Tokyo, Shinjuku-ku
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
- Mexico (4):
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - H. Central Dr Ignacio M. P., San Luis Potosí City
  - Centro Especializado en Terapia Endovascular (CETEN), Zapopan, Jalisco
- Netherlands (8):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Catharina Ziekenhuis, Eindhoven
  - Scheper Ziekenhuis, Emmen
  - Admiraal de Ruyter Ziekenhuis, Goes
  - UMCG, Groningen
  - St. Antonius ziekenhuis, locatie Nieuwegein, Nieuwegein
  - Canisius-Wilhelmina ziekenhuis, Nijmegen
  - Ziekenhuis Bernhoven Uden, Uden
- Waikato Hospital, Hamilton, New Zealand
- Norway (5):
  - Sørlandet sykehus HF, Avd. Arendal, Arendal
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Stavanger Helseforskning, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (10):
  - Univ. Clinic Hosp, Bialystok, Bialystok
  - 10.Military Clin.Hospital&Polyclinic, Bydgoszcz
  - Swissmed Vascular Sp. Z.o.o Hosp., Cardiology Dept., Gdansk, Gdansk
  - University Clinical Center, Gdansk, Gdansk
  - Reg.Hosp Kielce,Swietokrzyskie,1.Clinic of Cardiology,Kielce, Kielce
  - Independent Public Clin.Hosp.#4, Cardiology Clinic,Lubilin, Lublin
  - Independent Public Healthcare, Dept. of Cardiology, Pulawy, Puławy
  - Central Hospital of Medical Academy, Warsaw, Warsaw
  - Lower Silesian Spec.Hosp.T.Marciniaka,Cardiology Dep,Wroclaw, Wroclaw
  - John Paul II Regional Hospital, Zamosc, Zamość
- Portugal (7):
  - Hospital Garcia de Orta, EPE, Almada
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - Centro Hosp. de Leiria-Pombal, Leiria
  - CHLC, EPE - Hospital de Santa Marta, Lisbon
  - CHLO, EPE - Hospital de Santa Cruz, Lisbon
  - CHLN, EPE - Hospital de Santa Maria, Lisbon
  - CHUC,EPE - Hospital Geral dos Covões, S. Martinho Do Bispo,Coimbra
- Russia (14):
  - Altaiskyi Reg.Cardiologic Dispensary,Cardiology Dept,Barnaul, Barnaul
  - Regional Clinical Hospital No.3, Cardiology Dept,Chelyabinsk, Chelyabinsk
  - State Instit.Kazan Fed.Univ., Kazan'
  - State Autonomous Healthc Insti City Clin Hosp#7,Cardio,Kazan, Kazan'
  - Res.Inst.-Compl.Iss.Cardi.Dis., Kemerovo
  - Clin.Hosp.#1na S.V.Ochapovskiy, Krasnodar
  - City Clin.Hosp.#15 n.a.O.M.Filatov,Cardiology Dept.#2,Moscow, Moscow
  - City Clin.Hosp#51,Moscow Healthcare Dep.X-ray surgery method, Moscow
  - Cntr of CV Surgery na Bakulev,Surg.Treatm of Inter.Path.dept, Moscow
  - North-Western Fed.Med.Resear.Centr na V.I.Almazov,Cardio.dep, Saint Petersburg
  - City Pokrovskiy Hospital, Cardiology Dept., Saint Petersburg, Saint Petersburg
  - State Budg.Healthc.Instit.Samara Reg.Clin.Cardiology Dispens, Samara
  - State Budg.Healthc.Instit Volgograd RegClin.Cardiology Centr, Volgograd
  - Cent.f.Spec.Med.C.U.Cardi.Inst, Yekaterinburg
- Singapore (2):
  - National University Hospital, Singapore
  - National Heart Center, Singapore
- Slovakia (4):
  - Slov.Ins.Crdi.Dise.,Cor.C.U., Banská Bystrica
  - Nat.Instit.Cardiov.Diseas,Arryhythmias&Cardiac Pacing,Bratis, Bratislava
  - East Slovak Inst.Cardi.Disea., Košice
  - Kardiocentrum Nitra,Internal Medicine Dept, Nitra, Nitra
- Slovenia (4):
  - General Hospital Celje, Celje
  - General Hospital Izola, Cardiology Department, Izola
  - University Medical Center Ljubljana, Ljubljana
  - Univ. Medical Center Maribor, Maribor
- South Korea (13):
  - Inje University Haeundae Paik Hospital, Busan
  - Kyungpook National Univ. Hosp, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Pusan National Univ. Hosp, Pusan
  - Kyung Hee University Hospital, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Severance Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - St.Carollo Hospital, Suncheon
  - Ajou University Hospital, Suwon
  - Wonju Severance Christian Hosp, Wŏnju
- Spain (14):
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Bellvitge, L'Hospitalet Llobregat (bcn)
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - Hospital de Manises, Manises
  - Hospital Virgen de la Victoria, Málaga
  - CS Parc Taulí, Sabadell (Barcelona)
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Virgen del Rocío, Seville
  - Hospital de Galdakao, Vizcaya
  - Hospital Miguel Servet, Zaragoza
- Sweden (8):
  - Länssjukhuset, Gävle, Gävle
  - Sahlgrenska Universitetssjukhuset, Östra, Gothenburg
  - Länssjukhuset, Halmstad, Halmstad
  - Lasarettet, Helsingborg, Helsingborg
  - Universitetssjukhuset, Linköping, Linköping
  - Skånes universitetssjukhus, Lund, Lund
  - Skånes universitetssjukhus, Malmö, Malmo
  - Danderyds Sjukhus, Stockholm
- Taiwan (8):
  - Chang-Hua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - NCKUH, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan District
- Thailand (4):
  - Siriraj Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (16):
  - Cukurova Universitesi Tip Fakultesi Kardiyoloji AnabilimDali, Adana
  - Türkiye Yüksek Ihtisas Egitim ve Arastirma Hastanesi, Ankara
  - Diskapi Yildirim Beyazit EAH, Ankara
  - Bursa Yuksek Ihtisas EAH, Bursa
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Kardiyoloji Enstitusu, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - Bagcilar Egitim ve Arastirma Hastanesi, Istanbul
  - Medipol Mega Üniversitesi Hastanesi, Istanbul
  - Istanbul Mehmet Akif Ersoy Egitim ve Arastirma Hastanesi, Istanbul
  - Siyami Ersek Gogus Kalp ve Damar Cerrahisi Hastanesi, Istanbul
  - Kartal Kosuyolu Yuksek Ihtisas EAH, Istanbul
  - Dokuz Eylul Unv. Tip Fakultesi, Izmir
  - Izmir Katip Celebi Univ. EAH, Izmir
  - Erciyes Universitesi Tip Fakultesi Kardiyoloji Anabilim Dali, Kayseri
  - Ondokuz Mayis Universitesi Tip Fakultesi, Samsun
- United Kingdom (12):
  - Birmingham City Hospital, Birmingham
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Royal Derby Hospital, Derby
  - Dorset County Hospital, Dorchester
  - Grantham District Hospital, Grantham
  - Wycombe General Hospital, High Wycombe
  - Glenfield Hospital, Leicester
  - Lincoln County Hospital, Lincoln
  - St Bartholomew's Hospital, London
  - Altnagelvin Area Hospital, Londonderry
  - James Cook University Hospital, Middlesbrough
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Nicolau JC, Bhatt DL, Hohnloser SH, Kimura T, Lip GYH, Miede C, Nordaby M, Oldgren J, Steg PG, Ten Berg JM, Godoy LC, Cannon CP; RE-DUAL PCI Steering Committee and Investigators. Dabigatran Dual Therapy vs Warfarin Triple Therapy Post-Percutaneous Coronary Intervention in Patients with Atrial Fibrillation With/Without a Proton Pump Inhibitor: A Pre-Specified Analysis of the RE-DUAL PCI Trial. Drugs. 2020 Jul;80(10):995-1005. doi: 10.1007/s40265-020-01323-x. PMID 32562206
- [Derived] De Caterina R, Procopio A, Lopez Sendon JL, Raev D, Mehta SR, Opolski G, Oldgren J, Steg PG, Hohnloser SH, Lip GYH, Kimura T, Kleine E, Ten Berg JM, Bhatt DL, Miede C, Nordaby M, Cannon CP; RE-DUAL PCI Steering Committee and Investigators. Comparison of Dabigatran Plus a P2Y12 Inhibitor With Warfarin-Based Triple Therapy Across Body Mass Index in RE-DUAL PCI. Am J Med. 2020 Nov;133(11):1302-1312. doi: 10.1016/j.amjmed.2020.03.045. Epub 2020 May 7. PMID 32389658
- [Derived] Berry NC, Mauri L, Steg PG, Bhatt DL, Hohnloser SH, Nordaby M, Miede C, Kimura T, Lip GYH, Oldgren J, Ten Berg JM, Cannon CP. Effect of Lesion Complexity and Clinical Risk Factors on the Efficacy and Safety of Dabigatran Dual Therapy Versus Warfarin Triple Therapy in Atrial Fibrillation After Percutaneous Coronary Intervention: A Subgroup Analysis From the REDUAL PCI Trial. Circ Cardiovasc Interv. 2020 Apr;13(4):e008349. doi: 10.1161/CIRCINTERVENTIONS.119.008349. Epub 2020 Apr 7. PMID 32252548
- [Derived] Hohnloser SH, Steg PG, Oldgren J, Nickenig G, Kiss RG, Ongen Z, Navarro Estrada JL, Oude Ophuis T, Lip GYH, Nordaby M, Kleine E, Ten Berg JM, Bhatt DL, Cannon CP; RE-DUAL PCI Steering Committee and Investigators. Renal Function and Outcomes With Dabigatran Dual Antithrombotic Therapy in Atrial Fibrillation Patients After PCI. JACC Cardiovasc Interv. 2019 Aug 26;12(16):1553-1561. doi: 10.1016/j.jcin.2019.05.050. PMID 31439336
- [Derived] Chi G, Kerneis M, Kalayci A, Liu Y, Mehran R, Bode C, Halperin JL, Verheugt FWA, Wildgoose P, van Eickels M, Lip GYH, Cohen M, Peterson ED, Fox KAA, Gibson CM. Safety and efficacy of non-vitamin K oral anticoagulant for atrial fibrillation patients after percutaneous coronary intervention: A bivariate analysis of the PIONEER AF-PCI and RE-DUAL PCI trial. Am Heart J. 2018 Sep;203:17-24. doi: 10.1016/j.ahj.2018.06.003. Epub 2018 Jun 13. PMID 30015064
- [Derived] Cannon CP, Bhatt DL, Oldgren J, Lip GYH, Ellis SG, Kimura T, Maeng M, Merkely B, Zeymer U, Gropper S, Nordaby M, Kleine E, Harper R, Manassie J, Januzzi JL, Ten Berg JM, Steg PG, Hohnloser SH; RE-DUAL PCI Steering Committee and Investigators. Dual Antithrombotic Therapy with Dabigatran after PCI in Atrial Fibrillation. N Engl J Med. 2017 Oct 19;377(16):1513-1524. doi: 10.1056/NEJMoa1708454. Epub 2017 Aug 27. PMID 28844193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged ≥80 years in the United States of America (USA) were assigned to 110 milligram (mg) Dual antithrombotic therapy with dabigatran etexilate (DE-DAT), 150 mg DE-DAT, or warfarin. All other patients including aged ≥80 years (for Japan ≥70 years) outside of the USA were assigned to 110 mg DE-DAT or warfarin
Pre-assignment Details: All patients (Pts) were screened for eligibility to participate in trial. Pts attended sites to ensure that they met all implemented inclusion/exclusion criteria. Pts were not to be randomised to trial drug if any of specific entry criteria was violated. In this study, 2725 Pts were entered & randomised. 2678 Pts were treated.
Groups:
- Dabigatran Etexilate 110mg: Patients were orally administered Dabigatran Etexilate 110mg capsule twice daily (BID) for at least 6 months.
- Dabigatran Etexilate 150mg: Patients were orally administered Dabigatran Etexilate 150mg capsule twice daily (BID) for at least 6 months.
- Warfarin: Patients were orally administered warfarin 1 mg, 3 mg, or 5 mg tablets once daily for at least 6 months. The warfarin dose was titrated as needed to maintain the target International normalised ratio (INR) of 2.0 to 3.0 (2.0 to 2.6 for Japanese patients aged ≥70 years); 2.0 to 2.5 if feasible
Period: Overall Study
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin
Started | 981 (Started are the Randomised/entered patients.) | 763 (Started are the Randomised/entered patients.) | 981 (Started are the Randomised/entered patients.)
Completed | 886 | 703 | 849
Not Completed | 95 | 60 | 132
Not completed — Trial disease worsening | 7 | 5 | 1
Not completed — Other pre-existing disease worsening | 6 | 4 | 9
Not completed — Other Adverse Event (AE) | 52 | 32 | 49
Not completed — Protocol Violation | 2 | 4 | 1
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Consent withdrawn, not due to AE | 21 | 8 | 56
Not completed — Other than stated | 3 | 4 | 14

BASELINE CHARACTERISTICS:
Population: The anaysis set used was Full analysis set (FAS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Total
Number analyzed (Participants) | 981 | 763 | 981 | 2725
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the time of signing informed consent form is presented. Population: FAS
  Years | 71.5 (8.87) | 68.6 (7.65) | 71.7 (8.90) | 70.8 (8.66)
Age, Customized [Count of Participants; unit: Participants]
  <80: EU/ROW | 725 | 699 | 718 | 2142
  <80: USA | 54 | 53 | 61 | 168
  ≥80: EU/ROW | 189 | 3 | 192 | 384
  ≥80: USA | 13 | 8 | 10 | 31
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 253 | 171 | 231 | 655
    Male | 728 | 592 | 750 | 2070
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Hispanic or Latino | 70 | 46 | 59 | 175
    Not Hispanic or Latino | 903 | 700 | 904 | 2507
    Unknown or Not Reported | 8 | 17 | 18 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The details on Race has been provided Population: FAS
  Participants
    Asian | 116 | 79 | 125 | 320
    Black | 5 | 7 | 3 | 15
    White | 851 | 658 | 835 | 2344
    Other | 5 | 8 | 7 | 20
    Missing | 4 | 11 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to First Adjudicated ISTH MBE or CRNMBE
Description: Time to event analysis of patients with first adjudicated International Society of Thrombosis and Haemostasis (ISTH) Major Bleeding Event (MBE) or Clinically Relevant Non Major Bleeding Event (CRNMBE). The number of observed patients with adjudicated ISTH MBE or CRNMBE was reported.
  Full analysis set (FAS): All consenting patients randomised were analysed in the treatment group to which they were randomised regardless of whether they took trial medication. The start date of the observation period for this analysis set was the date of randomisation. Patients who discontinued trial medication were followed until the end of the trial.
  Patients who were lost to follow-up for vital status were censored for the primary endpoint at the time of their last known vital status.
  Intention to treat period: The observation period for these analysis was the so called 'intention to treat period'.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Groups:
- Warfarin (Excluding Elder Patients Outside USA): Patients were orally administered warfarin once daily. The warfarin dose was titrated as needed to maintain the target INR of 2.0 to 3.0 ; 2.0 to 2.5 if feasible. Elderly patients who were outside the USA were excluded.
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 151 | 154 | 264 | 196
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; A pre-defined hierarchical testing approach was used. This was the first step in hierarchy. The upper bound of the Wald confidence interval (CI) of the HR of Dabigatran Etexilate 110mg vs Warfarin (one-sided 97.5%) was compared with this noninferiority margin for the testing of non-inferiority; Test type: Non-Inferiority — All non-inferiority tests were based on a margin of 1.38; p < 0.0001, Regression, Cox — P values for noninferiority were calculated at a one-sided alpha level of 0.025; The Cox proportional hazard model is stratified by age, non-elderly vs elderly [<70 or >=70 in Japan and <80 or >=80 years old elsewhere]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.42 to 0.63] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); A pre-defined hierarchical testing approach was used. This was the second step in hierarchy. The upper bound of the Wald confidence interval (CI) of the HR of Dabigatran Etexilate 150mg vs Warfarin (one-sided 97.5%) was compared with this noninferiority margin for the testing of non-inferiority; Test type: Non-Inferiority — All non-inferiority tests were based on a margin of 1.38; p < .0001, Regression, Cox — P-values for non-inferiority were calculated at a one-sided alpha level of 0.025; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.88] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 3: Comparison: Dabigatran Etexilate 110mg vs Warfarin; A pre-defined hierarchical testing approach was used. This was the fourth step in hierarchy; Test type: Superiority; p < 0.001, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.42 to 0.63] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 4: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); A pre-defined hierarchical testing approach was used. This was the sixth step in hierarchy; Test type: Superiority; p = 0.0020, Regression, Cox — unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded; Wald 2-sided p-value from (unstratified) Cox proportional hazards model; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.58 to 0.88]; Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

2. Secondary Outcome: Time to Adjudicated Undetermined Cause of Death
Description: Time to event analysis of patients with adjudicated Undetermined cause of death. The number of observed patients with adjudicated Undetermined cause of death was reported.
  This is referred to a death not attributable to cardiovascular (CV) death or to a non-cardiovascular (non-CV) cause. Inability to classify the cause of death may have been due to lack of information (e.g. the only available information was "patient died") or when there was insufficient supporting information or detail to assign the cause of death.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 4 | 5 | 4 | 3
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.9862, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.25 to 3.95] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; p = 0.5277, Regression, Cox; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.38 to 6.64] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

3. Secondary Outcome: Time to Adjudicated Non-CV
Description: Time to event analysis of patients with adjudicated Non-cardiovascular (Non-CV). The number of observed patients with adjudicated Non-CV was reported.
  Non-CV death was defined as any death with a specific cause that was not thought to be CV. These were possible examples of non-CV causes of death: Pulmonary, Renal, Gastrointestinal, Hepatobiliary, Pancreatic Infection(included sepsis), Inflammatory (e.g. systemic inflammatory response syndrome) or immune (including autoimmune), Haemorrhage that was neither CV bleeding nor a stroke, Non-CV procedure or surgery, Trauma, Suicide, Non-prescription drug reaction or overdose, Prescription drug reaction or overdose, Neurological (non-CV), Malignancy, Other non-CV
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 14 | 4 | 13 | 8
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.8853, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.50 to 2.25] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.2380, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.15 to 1.61] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

4. Secondary Outcome: Time to Adjudicated CV
Description: Time to event analysis of patients with adjudicated Cardiovascular (CV) death. The number of observed patients with adjudicated Cardiovascular (CV) death was reported.
  CV death included death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, death due to CV procedures, death due to CV haemorrhage, and death due to other CV causes.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 37 | 21 | 31 | 24
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.5252, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.72 to 1.88] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.5670, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.47 to 1.51] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

5. Secondary Outcome: Time to Adjudicated All Cause Death
Description: Time to event analysis of patients with adjudicated all cause death. The number of observed patients with adjudicated all cause death was reported. All cause death is defined as the death from any cause included CV death, non-CV death, and undetermined cause of death.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 55 | 30 | 48 | 35
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.5579, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.76 to 1.65] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.4414, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.51 to 1.34] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

6. Secondary Outcome: Time to First Adjudicated MI
Description: Time to event analysis of patients with first adjudicated Myocardial Infarction (MI). The number of observed patients with adjudicated MI was reported
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 44 | 26 | 29 | 22
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other — Wald 2-sided p-value from (stratified) Cox proportional hazards model; p = 0.0861, Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.94 to 2.41] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.6144, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.66 to 2.04] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

7. Secondary Outcome: Time to First Adjudicated Stroke
Description: Time to event analysis of patients with first adjudicated Stroke. The number of observed patients with adjudicated Stroke was reported.
  Stroke was defined as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury as a result of haemorrhage or infarction
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 17 | 9 | 13 | 8
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.4803, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.63 to 2.67] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.8537, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.42 to 2.83] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

8. Secondary Outcome: Time to First Adjudicated SE
Description: Time to event analysis of patients with first adjudicated Systemic embolism (SE). The number of observed patients with adjudicated SE was reported.
  SE is an acute vascular occlusion of the extremities or any organ (kidneys, mesenteric arteries, spleen, retina or grafts) and had to be documented by angiography, surgery, scintigraphy, or autopsy.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 3 | 1 | 3 | 3
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.9388, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.19 to 4.66] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.3030, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.03 to 2.93] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

9. Secondary Outcome: Time to First Adjudicated ST
Description: Time to event analysis of patients with first adjudicated Stent Thrombosis (ST). The number of observed patients with adjudicated ST was reported.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 15 | 7 | 8 | 7
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.1546, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.86, 95% CI 2-sided [0.79 to 4.40] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.9789, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.35 to 2.81] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

10. Secondary Outcome: Time to Composite Endpoint of Death + MI + Stroke
Description: Time to event analysis of patients with the composite endpoint of death + myocardial infarction (MI) + stroke. The number of observed patients with the composite endpoint of death + myocardial infarction (MI) + stroke was reported.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 107 | 60 | 80 | 57
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.0484, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [1.00 to 1.79] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.8903, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.71 to 1.47] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

11. Secondary Outcome: Time to Composite Endpoint of Death or First Thrombotic Event
Description: Time to event analysis of patients with composite endpoint of death or first thrombotic event (all death, myocardial infarction (MI), stroke/systemic embolism (SE)). The number of observed patients with composite endpoint of death or thrombotic event (all death, MI, stroke/SE).
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Groups:
- Warfarin (Excluding Elder Patients Outside USA: Patients were orally administered warfarin once daily. The warfarin dose was titrated as needed to maintain the target INR of 2.0 to 3.0 ; 2.0 to 2.5 if feasible. Elderly patients who were outside the USA were excluded.
- All Dabigatran Etexilate: Patients in combined Dabigatran Etexilate group (ie 110 mg DE + 150 mg DE).
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA | All Dabigatran Etexilate
Number analyzed (Participants) | 981 | 763 | 981 | 764 | 1744
Participants | 108 | 60 | 83 | 60 | 168
Statistical Analysis 1: Comparison: Warfarin vs All Dabigatran Etexilate; A pre-defined hierarchical testing approach was used. This was the fifth step in hierarchy; Test type: Non-Inferiority — All non-inferiority tests were based on a margin of 1.38; p = 0.1128, Regression, Cox — P values for noninferiority were calculated at a one-sided alpha level of 0.025; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.90 to 1.53] — The upper bound of the Wald confidence interval (CI) of the HR of All Dabigatran Etexilate (110mg and 150 mg) vs Warfarin (one-sided 97.5%) was compared with this noninferiority margin for the testing of non-inferiority
Statistical Analysis 2: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.0720, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.98 to 1.73] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 3: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA; Test type: Other; p = 0.8750, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.68 to 1.39] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

12. Secondary Outcome: Time to First Adjudicated Unplanned Revascularisation by PCI/CABG
Description: Time to event analysis of patients with adjudicated unplanned revascularisation by Percutaneous Coronary Intervention (PCI)/Coronary Artery Bypass Graft (CABG). The number of observed patients with adjudicated unplanned revascularisation by PCI/CABG was reported.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA)
Number analyzed (Participants) | 981 | 763 | 981 | 764
Participants | 76 | 51 | 69 | 52
Statistical Analysis 1: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.6080, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.79 to 1.51] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 2: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.8348, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded from; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.65 to 1.41] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

13. Secondary Outcome: Time to Death or First Thrombotic Event or Unplanned Revascularisation by PCI/CABG
Description: Time to event analysis of patients with death or thrombotic event (all death, myocardial infarction, stroke/systemic embolism) or unplanned revascularisation by Percutaneous Coronary Intervention/Coronary Artery Bypass Graft. The number of observed patients with death or first thrombotic event or unplanned revascularisation by PCI/CABG was reported.
Time Frame: up to 30 months
Population: Full Analysis set (FAS) following the intention-to-treat principle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin | Warfarin (Excluding Elder Patients Outside USA) | All Dabigatran Etexilate
Number analyzed (Participants) | 981 | 763 | 981 | 764 | 1744
Participants | 149 | 90 | 131 | 98 | 239
Statistical Analysis 1: Comparison: Warfarin vs All Dabigatran Etexilate; A pre-defined hierarchical testing approach was used. This was the third step in hierarchy; Test type: Non-Inferiority — All non-inferiority tests were based on a margin of 1.38; p = 0.0047, Regression, Cox — P values for noninferiority were calculated at a one-sided alpha level of 0.025; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.84 to 1.29] — [estimate comment as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Dabigatran Etexilate 110mg vs Warfarin; Test type: Other; p = 0.3002, Regression, Cox — Wald 2-sided p-value from (stratified) Cox proportional hazards model; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.90 to 1.43] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model
Statistical Analysis 3: Comparison: Dabigatran Etexilate 150mg vs Warfarin (Excluding Elder Patients Outside USA); Test type: Other; p = 0.4432, Regression, Cox — Wald 2-sided p-value from (unstratified) Cox proportional hazards model; unstratified Cox proportional hazards model was used and elderly patients outside the USA were excluded; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.67 to 1.19] — Hazard Ratio (HR) and Wald confidence intervals are derived from a Cox proportional-hazard model

ADVERSE EVENTS:
Time Frame: From the first intake of randomised trial drug until 6 days after the last intake of the randomised trial drug, ie., up to 31 Months.
Description: Treated set (TS): The set of patients who received at least 1 dose of trial medication was analysed according to the treatment they had received. The start date of the observation period for this analysis set was the date of the first intake of trial medication.
  All on-treatement AE's for this study were reported based on the Treated set
Arm/Group | Dabigatran Etexilate 110mg | Dabigatran Etexilate 150mg | Warfarin
All-Cause Mortality (participants affected / at risk) | 38/972 | 24/758 | 41/948
Serious Adverse Events (participants affected / at risk) | 415/972 | 300/758 | 396/948
Other Adverse Events (participants affected / at risk) | 128/972 | 126/758 | 229/948
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 110mg (N=972) | Dabigatran Etexilate 150mg (N=758) | Warfarin (N=948)
Anaemia (Blood and lymphatic system disorders) | 6 | 7 | 7
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 2 | 4
Acute left ventricular failure (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 20 | 14 | 15
Acute right ventricular failure (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 20 | 18 | 18
Angina unstable (Cardiac disorders) | 26 | 15 | 13
Aortic valve disease (Cardiac disorders) | 0 | 0 | 1
Aortic valve disease mixed (Cardiac disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 2 | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 44 | 36 | 34
Atrial flutter (Cardiac disorders) | 18 | 8 | 6
Atrial tachycardia (Cardiac disorders) | 1 | 1 | 0
Atrial thrombosis (Cardiac disorders) | 2 | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 0 | 1 | 1
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 5 | 5 | 6
Cardiac arrest (Cardiac disorders) | 4 | 1 | 5
Cardiac asthma (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 48 | 30 | 46
Cardiac failure acute (Cardiac disorders) | 7 | 5 | 4
Cardiac failure chronic (Cardiac disorders) | 7 | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 14 | 13 | 19
Cardiac flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 6 | 6 | 7
Coronary artery insufficiency (Cardiac disorders) | 0 | 1 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 4 | 12 | 3
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 2 | 0
Left ventricular failure (Cardiac disorders) | 3 | 0 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 5 | 0 | 3
Mitral valve prolapse (Cardiac disorders) | 0 | 1 | 0
Myocardial fibrosis (Cardiac disorders) | 0 | 2 | 0
Myocardial infarction (Cardiac disorders) | 17 | 8 | 8
Myocardial ischaemia (Cardiac disorders) | 3 | 1 | 5
Palpitations (Cardiac disorders) | 1 | 0 | 2
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Pericarditis constrictive (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 0 | 1 | 3
Silent myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 5 | 2 | 3
Supraventricular tachycardia (Cardiac disorders) | 1 | 1 | 0
Systolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 2 | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 5 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1
Trifascicular block (Cardiac disorders) | 0 | 1 | 0
Ventricle rupture (Cardiac disorders) | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 7 | 5 | 3
Generalised resistance to thyroid hormone (Congenital, familial and genetic disorders) | 0 | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Venous angioma of brain (Congenital, familial and genetic disorders) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 1
Thyroid mass (Endocrine disorders) | 1 | 0 | 0
Blindness transient (Eye disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 2 | 3 | 3
Eye haemorrhage (Eye disorders) | 0 | 1 | 1
Glaucoma (Eye disorders) | 3 | 2 | 2
Neovascular age-related macular degeneration (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 3
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 2
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 5 | 13
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 3 | 2
Hiatus hernia (Gastrointestinal disorders) | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 3
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 2
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 4 | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 4 | 3 | 4
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Stomach mass (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 5
Cardiac death (General disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 3 | 1 | 0
Chest pain (General disorders) | 14 | 15 | 15
Death (General disorders) | 8 | 6 | 5
Device related thrombosis (General disorders) | 1 | 0 | 0
Drug effect increased (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1
Impaired healing (General disorders) | 2 | 1 | 1
Implant site haematoma (General disorders) | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0
Medical device site haematoma (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 3 | 3 | 1
Oedema (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 1
Sudden cardiac death (General disorders) | 4 | 2 | 1
Sudden death (General disorders) | 2 | 1 | 7
Ulcer (General disorders) | 1 | 1 | 0
Ulcer haemorrhage (General disorders) | 0 | 1 | 0
Vascular stent occlusion (General disorders) | 0 | 1 | 0
Vascular stent restenosis (General disorders) | 5 | 4 | 3
Vascular stent stenosis (General disorders) | 1 | 0 | 0
Vascular stent thrombosis (General disorders) | 25 | 10 | 17
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 4 | 2 | 4
Cholecystitis acute (Hepatobiliary disorders) | 2 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 4 | 1 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 2
Candida infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 6 | 3
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 2 | 0 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 1 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 1
Endocarditis (Infections and infestations) | 2 | 1 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 2 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 0 | 1 | 0
Gangrene (Infections and infestations) | 2 | 2 | 0
Gastritis viral (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Hepatitis C (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 1 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 3 | 3
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 2 | 1
Orchitis (Infections and infestations) | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 3 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 20 | 15 | 19
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 2 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 2 | 0 | 1
Sepsis (Infections and infestations) | 5 | 5 | 4
Septic shock (Infections and infestations) | 0 | 3 | 2
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Systemic infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 3 | 4
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 3 | 0 | 1
Vestibular neuronitis (Infections and infestations) | 2 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Chemical burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Confusion postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 2 | 5
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 2
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 2
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Splenic injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 3
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood pressure abnormal (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 1
Blood urine (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Haematocrit decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 4 | 2
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 9
Liver function test increased (Investigations) | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 2
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 4 | 2
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plica syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 4
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 3
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Rectal cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Urinary bladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 0 | 1
Basal ganglia stroke (Nervous system disorders) | 1 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 1 | 1
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 0 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 3 | 4 | 4
Dementia (Nervous system disorders) | 3 | 1 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 3
Dizziness postural (Nervous system disorders) | 0 | 0 | 1
Drop attacks (Nervous system disorders) | 0 | 0 | 1
Encephalomalacia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 3 | 0
Hemiplegia (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 4 | 4 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0
Lateral medullary syndrome (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Mental impairment (Nervous system disorders) | 1 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 0 | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0
Quadriparesis (Nervous system disorders) | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Spinal claudication (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 9 | 10 | 7
Tension headache (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 4 | 1 | 1
Device malfunction (Product Issues) | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 2
Delirium (Psychiatric disorders) | 3 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Transient psychosis (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 15 | 14 | 6
Acute prerenal failure (Renal and urinary disorders) | 0 | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 3 | 4 | 7
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 3 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 3 | 2
Renal impairment (Renal and urinary disorders) | 3 | 1 | 1
Renal infarct (Renal and urinary disorders) | 0 | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 6
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 17
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0 | 0
Angiodysplasia (Vascular disorders) | 1 | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 2 | 1
Aortic dissection (Vascular disorders) | 1 | 0 | 0
Aortic dissection rupture (Vascular disorders) | 1 | 0 | 0
Aortic necrosis (Vascular disorders) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 3 | 0 | 2
Aortic thrombosis (Vascular disorders) | 0 | 0 | 1
Aortitis (Vascular disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1 | 1
Diabetic vascular disorder (Vascular disorders) | 0 | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 1
Femoral artery dissection (Vascular disorders) | 0 | 0 | 1
Haematoma (Vascular disorders) | 2 | 1 | 7
Haemorrhage (Vascular disorders) | 2 | 2 | 6
Hypertension (Vascular disorders) | 6 | 5 | 1
Hypertensive crisis (Vascular disorders) | 8 | 3 | 11
Hypertensive emergency (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 6
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 1 | 1 | 0
Ischaemia (Vascular disorders) | 1 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 5 | 1 | 5
Peripheral artery occlusion (Vascular disorders) | 0 | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 0 | 1
Peripheral embolism (Vascular disorders) | 2 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 2 | 0
Shock (Vascular disorders) | 0 | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 2 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran Etexilate 110mg (N=972) | Dabigatran Etexilate 150mg (N=758) | Warfarin (N=948)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 62 | 60 | 61
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 52 | 59 | 146
Haematoma (Vascular disorders) | 27 | 24 | 60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02164864/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT02164864/SAP_001.pdf